CLINICAL TRIAL: NCT01647867
Title: Study of the Expression of Met Receptor Fragments in Non Small Cell Lung Cancers
Acronym: MetLung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MetLung - 1204
Record Dates: First submitted 2012-07-17; First posted 2012-07-24 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Met fragments expression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Met analysis (Experimental): Met analysis on tissue and blood Western Blot Immunohistochemistry ELISA test
  Interventions: Other: Met analysis on tissue and blood

INTERVENTIONS:
Other: Met analysis on tissue and blood — 10 mL of blood and 4 pieces of tissue (2 of tumor tissue, 2 of healthy tissue) all taken at the same time as surgery or bronchoscopy, depending on the stage of the disease

SUMMARY:
Our project, established through collaboration between clinicians (Oscar Lambret Center-University Hospital) and scientists (IBL), aims to evaluate the expression of Met fragments in the lung cancer (LC). Unlike previous studies on Met by sequencing, in situ hybridization or immunohistochemistry, the investigators propose a protein analysis by Western blot of tumor samples and healthy tissue. This approach will evaluate the expression of full-length receptor, the potential presence of intracellular fragments, and their phosphorylation status.

DETAILED DESCRIPTION:
* Patient information and collection of signed inform consent
* Blood sample collection before bronchoscopy or before surgery, at the same time as a usual blood assessment.
* Prospective collection of bronchial biopsies of patients with metastatic non small cell lung cancer, during a bronchoscopy at the Oscar Lambret Center (Dr Dansin)
* Prospective collection of resected specimens of patients with localized non small cell lung cancer, who were operated at the thoracic surgery unit of the University hospital (Pr Porte)
* Transportation of the samples to the pathology laboratories (Dr Robin, Pr Copin)
* Selection of blocks of interest and preparation of tumor samples
* Clinical data collection : date of biopsy or surgery, disease-free survival, overall survival, tumor characteristics, EGFR status, ALK, BRAF, HER2
* Transportation of tumor blocks and blood samples to the Institute of Biology of Lille for analyses: Western blot, immunohistochemistry and ELISA test)
* Return to storage of the tumor samples at the Oscar Lambret Center and at the University hospital of Lille

ELIGIBILITY:
Inclusion Criteria:

* Patients with non small cell lung cancer (NSCLC)
* Patients candidate for bronchial biopsies at the Oscar Lambret Center (metastatic stage) or candidate for thoracic surgery at University Hospital of Lille (localized stage)
* Treatment naive patient for metastatic NSCLC
* Patients with or without neoadjuvant therapy for localized NSCLC
* Male or female patients aged ≥ 18 years
* Patient registered with the social security system
* Having signed a written Informed Consent

Exclusion Criteria:

* Malignant tumors which are not carcinoma
* Small-cell malignant tumors
* Secondary bronchial lesions
* Revision surgery
* Pregnant or breastfeeding women
* Patient under guardianship or tutorship
* Previous cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Expression and localization of Met C-terminal active fragments in NSCLC | baseline
  Western Blot and immunohistochemistry

SECONDARY OUTCOMES:
Evaluation of the activation of Met receptor | baseline
  Activation of Met receptor by immunochemical analysis (Western Blot)
Correlation between expression of Met receptor fragments with clinical characteristics and/or prognosis factors as sex, TNM, EGFR status, histology, smoking status, survival | baseline
  Relationships between Met receptor expression and sex, TNM, EGFR status, histology, smoking status, survival
Expression in plasma of N-terminal Met fragments | baseline
  ELISA test

CONTACTS AND LOCATIONS:
Overall Officials: Eric DANSIN, MD, Study Director — Centre Oscar Lambret; David TULASNE, PhD, Study Director — Institute of Biology of Lille
Locations (2):
- France (2):
  - Centre Hospitalier Régional et Universitaire, Lille
  - Oscar Lambret Center, Lille

IPD SHARING:
Plan to Share IPD: No